CLINICAL TRIAL: NCT03613168
Title: The Pilot Study of Trastuzumab in Combination With Gemcitabine Plus Cisplatin for HER2-positive Biliary Tract Cancer
Brief Title: Trastuzumab in HER2-positive Biliary Tract Cancer
Acronym: BILHER
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Changhoon Yoo (Other)
Responsible Party: Sponsor-Investigator, Changhoon Yoo, Assistant professor, Asan Medical Center
Organization: Asan Medical Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BTC-HER2
Record Dates: First submitted 2018-07-28; First posted 2018-08-02 (Actual); Last update posted 2021-01-05 (Actual); Status verified 2021-01

CONDITIONS: Cholangiocarcinoma; Biliary Tract Cancer; HER-2 Protein Overexpression; HER-2 Gene Amplification
Keywords: Cholangiocarcinoma; Biliary Tract Cancer; Trastuzumab
MeSH Terms: conditions — Cholangiocarcinoma; Biliary Tract Neoplasms | interventions — Trastuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Trastuzumab plus Gem/Cis (Experimental): Gemcitabine 1,000 mg/m2 Day 1 and Day 8, every 3 weeks Cisplatin 25 mg/m2 Day 1 and Day 8, every 3 weeks Trastuzumab, every 3 weeks, 8 mg/kg at first cycle then, 6 mg/kg
  Interventions: Drug: Trastuzumab

INTERVENTIONS:
Drug: Trastuzumab — Trastuzumab plus gemcitabine/cisplatin

SUMMARY:
Trastuzumab is approved for the treatment of HER2-positive breast cancer and gastric cancer. The recent study showed that HER2 overexpression or amplification is noted about 5-15% of total biliary tract cancer patients. The aim of this study is to evaluate the efficacy and safety of trastuzumab in the combination of current standard gemcitabine plus cisplatin.

ELIGIBILITY:
Inclusion Criteria:

1. The subject with disease that is not amendable to a curative treatment approach or locally advanced or metastatic or unresectable CCC with histological diagnosis
2. At least one measurable(per RECIST 1.1) lesion
3. Primary or metastatic tumor with HER2 positive defined on IHC2+, FISH+ or IHC3+
4. ECOG Performance status 0 or 1
5. At least 3 months for life expectancy Common inclusion criteria
6. Men or women over 19 years at time of signing ICF
7. Signed Informed Consent Form

   Exclusion Criteria:
8. Received prior chemotherapy for advanced/metastatic disease (the adjuvant/neoadjuvant chemotherapy completed at least 6 months before enrolled will be accepted)
9. Not recovery from toxicities related to any prior treatments excluding alopecia (eg, neurological toxicity to ≥ Grade 2)
10. History of malignancy other than CCC within 5 years prior to screening, with the exception of malignancies with a negligible risk of metastasis or death, such as carcinoma in situ or thyroid papillary carcinoma Hematology, chemistry or organ function
11. ANC < 1.5 × 109/L, or Platelet < 100 × 109/L
12. Total bilirubin > 1.5 × ULN; or AST/ ALT > 2.5 × ULN (or if the tumor has expanded into the liver, > 5 × ULN); or, alkaline phosphatase > 2.5 × ULN (or > 5 × if the tumor has expanded into the liver, or > 10 × ULN if the tumor has expanded into the brain without liver,); or albumin < 2.5 g/dL
13. Creatinine clearance < 60 mL/min(calculated using the Cockcroft-Gault formula) Other exclusion criteria related to IP
14. History of proved congestive heart failure; angina with medication; evidence of transmural myocardial infarction on ECG; uncontrolled hypertension(systolic> 180 mmHg or diastolic> 100 mmHg); clinically significant heart valve disease; uncontrolled arrhythmia
15. LVEF < 50% (calculated by cardiac sonography or MUGA)
16. Subject with rest dyspnea due to metastatic tumor or other disease or who needs oxygen therapy
17. Chronic or high-dose corticosteroid treatment
18. Clinically significant Hearing impairment Common exclusion criteria
19. History or evidence of CNS metastases
20. Interstitial pneumonia or pulmonary fibrosis with symptom and exact lesion on chest X-ray
21. Hearing loss
22. Uncontrolled significant systemic disease (eg, infection or uncontrolled DM)
23. Pregnant or lactating females
24. Sexually active fertile subjects without contraception
25. Treatment with other investigational therapy within 4 weeks prior to initiation of study treatment
26. Radiotherapy within 4 weeks prior to initiation of study treatment (the rest at least 2 weeks after palliative radiotherapy for bone metastasis and recovery from the effects of radiation will be accepted.)
27. Major surgery within 4 weeks prior to initiation of study treatment
28. History of HIV and active HBV or HCV
29. Previously identified allergy or hypersensitivity to components of the study treatment formulations

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2020-11-01 (Actual); Study Completion 2021-01-04 (Actual)

PRIMARY OUTCOMES:
Response rate | 6 months
  Best response according to the Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1
Adverse events | 2 years
  Adverse events graded by National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) version 4.03

SECONDARY OUTCOMES:
Progression-free survival | 2 years
  Time between the initiation of chemotherapy and disease progression or death
Overall survival | 2 years
  Time between the initiation of chemotherapy and any cause of death

CONTACTS AND LOCATIONS:
Overall Officials: Changhoon Yoo, MD, Principal Investigator — Asan Medical Center
Locations (1):
- Asan Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No